CLINICAL TRIAL: NCT05884294
Title: Midline Catheter Versus Long Peripheral Intravenous Catheter in Hospitalized Adult Patients: Randomized Clinical Trial With Economic Analysis From the Perspective of the Public Health System.
Brief Title: Midline Catheter Versus Long Peripheral Intravenous Catheter in Hospitalized Adult Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022-0363
Record Dates: First submitted 2023-01-27; First posted 2023-06-01 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Vascular Access Devices
Keywords: vascular access device; midline catheter; long Peripheral Intravenous Catheter

STUDY DESIGN:
Intervention Model Description: randomized, parallel, open, controlled, and single-center clinical trial.
Who Masked: Outcomes Assessor
Masking Description: This study will be blind to statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PowerGlide Pro Midline catheter. (Experimental): The Intervention Group will be represented by hospitalized adult clinical patients who have been identified with difficult intravenous access. These patients will receive an ultrasound-guided insertion of the PowerGlide ProTM Midline 20G (10 cm).
  Interventions: Device: PowerGlide Pro Midline catheter.
- Introcan Safety Deep Access long peripheral venous catheter. (No Intervention): The control group will be subjected to the same selection criteria as the patients in the intervention group; however, they will receive an ultrasound-guided insertion of a long peripheral venous catheter Introcan Safety Deep Access 20G (6.4 cm).

INTERVENTIONS:
Device: PowerGlide Pro Midline catheter. — The Intervention Group will be represented by hospitalized adult clinical patients who have been identified with difficult intravenous access. These patients will receive an ultrasound-guided insertion of the PowerGlide ProTM Midline 20G (10 cm).
  Arms: PowerGlide Pro Midline catheter.

SUMMARY:
This research seeks to compare two types of vascular access (catheters that are inserted into the vein) for patient treatment during hospitalization. This research will evaluate how long each catheter lasts before presenting problems that may lead to its removal from the vein (the most common are swelling on the site of the catheter, clogging of the catheter, infections, or other less common problems. Each patient will be randomly selected to receive either catheter. In this study, we will also estimate how much each patient will spend if any of the problems mentioned occur.

DETAILED DESCRIPTION:
This randomized, parallel, open, controlled, single-center clinical trial is blind to outcome analysis. The use of midline catheter will be compared, regarding duration of use without complications, to the use of long peripheral intravenous catheter during continuous our intermittent intravenous therapy in adult clinical patients who have been hospitalized for up to 30 days. The intervention group will consist of hospitalized adult clinical patients who were identified with difficult intravenous access (DIVA) and who received medical indication of continuous or intermittent intravenous therapy for more than five and a maximum of 30 days of treatment. These patients will receive PowerGlide ProTM Midline catheter. The control group will consist of patients with the same profile described as the intervention group and will receive the insertion of a long peripheral venous catheter Introcan Safety Deep Access. At the end of the study, an economic analysis will be carried out from the perspective of the public health system if the intervention group shows favorable results.

ELIGIBILITY:
* patients hospitalized in a clinical ward unit;
* indicated for continuous or intermittent intravenous therapy more than five days;
* identified with difficult intravenous access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Lenght of time of vascular access without isolated or combined complications. | up to 30 days, end of therapy or withdrawal due to any complication
  Time in days.

SECONDARY OUTCOMES:
First-attempt puncture success | up to 30 days or end of therapy
  success in the first venipuncture, number venipuncture.

OTHER OUTCOMES:
Economic analysis | 30 days or end of therapy.
  micro-costing

CONTACTS AND LOCATIONS:
Overall Officials: Eneida R Rabelo da Silva, ScD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teixeira TO, Hansel LA, Ceratti RDN, Brum ID, Fernandes AGDS, Saline CG, Junges M, Rabelo-Silva ER. Midline catheter (10 cm) versus long peripheral intravenous catheter (6.4 cm): Randomized clinical trial protocol with economic analysis. PLoS One. 2025 Apr 24;20(4):e0319587. doi: 10.1371/journal.pone.0319587. eCollection 2025. PMID 40273075